CLINICAL TRIAL: NCT04057872
Title: PILOT STUDY in the Use of Therapeutic Plasma Exchange in Adult Patients With Severe Sepsis
Brief Title: Therapeutic Plasma Exchange in Adult Patients With Severe Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Responsible Party: Principal Investigator, Dr. George Alvarez, Intensivist, Department of Critical Care Medicine, Alberta Health Services, Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB19-1157
Record Dates: First submitted 2019-08-02; First posted 2019-08-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock
Keywords: Therapeutic Plasma Exchange (TPE); Septic Shock; Severe Sepsis; Albumin; Fresh Frozen Plasma
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Consecutive Adults patients with vasoplegic septic shock with at least 2 organ dysfunction will receive TPE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPE in Septic Shock (Experimental): The patients will undergo a dosing trial to determine safety and the most effective dose
  Interventions: Procedure: Therapeutic plasma exchange

INTERVENTIONS:
Procedure: Therapeutic plasma exchange — The removed plasma is 'exchanged or replaced' with either IV fluids, albumin, and/or Fresh frozen plasma

SUMMARY:
The incidence of sepsis (severe infection) has increased over the last four decades. Severe sepsis and septic shock are among the leading causes of death for patients admitted to critical care units with mortality ranging from 20-70% depending on totality of organ dysfunction. Outside of antibiotics and good bedside care, little has changed in the management of this life-threatening problem.

Therapeutic plasma exchange (TPE) involves the separation of plasma from whole blood. The removed plasma is 'exchanged or replaced' with either IV fluids, albumin, blood products or a combination thereof.

The primary objective of this study is to evaluate the safety of the TPE intervention protocol within 24 hours of study criteria being met. TPE is now a well-established program at the South Health Campus for neuro-muscular disorders. Since starting in May 2018, the investigators have performed over 150 runs making the SHC ICU one of the most experienced centers in Canada.

DETAILED DESCRIPTION:
Background

The incidence of sepsis has increased over the last four decades (1). Sepsis is a life-threatening condition that arises when the body's response to an infection injures its own tissues and organs. Severe sepsis and septic shock are among the leading causes of death for patients admitted to critical care units with mortality ranging from 20-70% depending on totality of organ dysfunction (2, 3). The literature is replete with initial promising phase 2 therapies failing in definitive randomized trails (4-8). In fact, a recent systematic review concluded that no evidence exists for any pharmacologic intervention that has consistently reduced mortality in critically ill patients (9). This is both surprising and frustrating for the author. The most recent guidelines have tried to redefine sepsis as a 'syndrome' since neither validated criterion nor do standard diagnostic tests exist (10). The authors argue that sepsis should be viewed as organ dysfunction caused by a dysregulated or non-homeostatic host response. Most of the clinical manifestations of severe infections are caused by an intense, generalized inflammatory response in the host mediated by a multitude of interrelated cellular and humoral factors (3).

Plasmapheresis or therapeutic plasma exchange (TPE) involves the separation of plasma from whole blood. The removed plasma is 'exchanged or replaced' with crystalloids, albumin, fresh frozen plasma or a combination thereof. TPE use is well established in many neurological disorders including Guillain-Barre syndrome (11), Myasthenia Gravis (12, 13) and antibody mediated syndromes(14, 15). It is considered the standard of care for thrombotic thrombocytopenic purpura (TTP) (16, 17). The rationale for the use of TPE in sepsis, a non-selective intervention, is to remove multiple toxic mediators including endotoxins, activated complement, pro-inflammatory cytokines and pro-coagulant factors (18, 19). If fresh-frozen plasma is used as replacement fluid, consumed plasma factors are substituted, thereby possibly restoring the opsonic capacity and improving the coagulation abnormalities and microcirculation.

Plasma exchange has been reported since the late 1970s as a potential adjunctive or salvage therapy in severe sepsis in both pediatric and adult patients (20-24). These case reports, retrospective reviews and observational studies suggest a survival advantage when compared to historical controls. However, the obvious bias limits any meaningful interpretation. A literature review found only 4 studies with any attempt at randomization. One study enrolled only adults (25), two were exclusively pediatric patients (26, 27) and one study involved both adults and children (28). Excluding the pediatric studies, the adult protocols had few similarities:

1. Reeves and colleagues attempted a multi-center Australian study but terminated enrollment after 22 adult and 8 children (28). The mean APACHEII scores for adults were 25.2. They aggressively exchanged 5 plasma volumes continuously over 36 hours using a combination of fresh frozen plasma (FFP) and albumin (1/4 ratio). Mortality was reported at 14 days. No data on ICU or hospital length of stay was provided. This trial reported significant decrease in certain inflammatory markers.
2. Busund's larger trail involved 106 adults and reported mortality at 28 days (25). They performed a single 30-40mls/kg exchange that could be repeated once if no clinical improvement was observed. The replacement used was FFP and albumin in a 1:1 ratio. Six episodes of transient hypotension and 1 allergic reaction to FFP was reported (the only trial to report adverse events). There was an encouraging trend towards improved survival (33% vs 53%) versus historical controls. No data on ICU or hospital length of stay was provided.

A more recent German pilot study tried to evaluate the safety and feasibility of enrollment within 12 hours of shock for a proposed randomized controlled trial (RCT) (29). The inclusion criteria were simple: (a) Current sepsis-3 definitions; noradrenaline dose >0.4ug/kg/min despite >30mls/kg of crystalloid; (b) Less than 12 hours of vasopressor support. They performed a single 1.2x plasma exchange using entirely FFP. The major findings were significantly less vasopressor support, fluid balance and a decline in plasma concentrations of pro-inflammatory mediators. The "sustained -responders" mortality was 43% vs 77% of non-responders, but the small numbers prevented statistical significance.

The use of plasma exchange in severe sepsis is graded by the American Society for Apheresis as category III with grade 2C indications, indicating that there is a lack of reliable trials to support TPE use in the condition (30). The purpose of this phase 1 clinical trial is to assess the safety of using plasma exchange in critically ill adult patients with septic shock. TPE is now a well-established program at the South Health Campus (SHC) for neuro-muscular disorders. Since starting in May 2018, we have performed over 240 runs in 43 patients making the SHC ICU the most experienced TPE center in Canada in the past 2 years. One plasma volume is currently the standard dose used safely in patients with neuro-muscular disorders at SHC.

Justification of Research

1. The incidence of sepsis has increased over 4 decades but no single pharmacological invention reduces mortality/morbidity.
2. A potential treatment that increases the chance of survival and recovery in patients with septic shock would be both beneficial to patients and help decrease medical costs from long term stays in the ICU.
3. The maximum tolerable dose of TPE in septic patients is unknown.

Study Objectives

Primary Objective: To evaluate the safety of the TPE intervention protocol within 24 hours of study criteria being met.

Secondary Objectives:

1. To evaluate preliminary efficacy of the TPE protocol.
2. To determine maximum tolerable dose of TPE in septic patients.
3. To record adverse events from TPE intervention.

Hypothesis

It is hypothesized that TPE will be safe for use in patients with septic shock. We will determine the maximum tolerable dose via a dose escalation study.

ELIGIBILITY:
Inclusion Criteria Adult patients (age ≥18) with a documented or strong clinical suspicion of infection that meets the definition of septic shock as per the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).

Exhibiting two of the four clinical signs of inflammation:

1. Core temperature > 38oC or < 36oC
2. Heart rate > 90 beats per minute
3. Respiratory rate > 20 breaths per minute, or PaCO2 < 32 mmHg, or mechanical ventilation
4. White cell count > 12 x 109/L or < 4 x 109/L or > 10% immature neutrophils

We will further identify the subset with a hospital mortality in excess of 40%:

1. >30 mls/kg fluid resuscitation
2. Noradrenaline >0.1 ug/kg/min to maintain MAP> 65mmHg for at least 4 consecutive hours and present at initiation of TPE
3. Lactate >2 mmol/l.

Exclusion Criteria Patients will be excluded in cases where death is deemed inevitable or imminent during admission and either the attending physician, patient or surrogate legal decision maker is not committed to active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | During course of ICU stay, could be up to 6 months
  Proportion of patients who experience at least 1 Adverse Event (AE)
Discontinue TPE | During course of ICU stay, could be up to 6 months
  Proportion of patients who discontinue TPE administration due to an AE
Enrollment Rate | During course of ICU stay, could be up to 6 months
  3. Enrollment rate (patients screened, patients eligible, patients approached, patients enrolled)
Protocol Completion | During course of ICU stay, could be up to 6 months
  Protocol completion (patients who complete study protocol)

SECONDARY OUTCOMES:
Organ dysfunction | During course of ICU stay, could be up to 6 months
  Resolution or worsening of organ dysfunction as per SOFA score
Vasopressor support | During course of ICU stay, could be up to 6 months
  Hours of vasopressor support
Ventilator support | During course of ICU stay, could be up to 6 months
  Days on ventilator if applicable
Days in ICU | During course of ICU stay, could be up to 6 months
  Days in ICU (censored to day ready for discharge)
Mortality | During course of ICU stay, could be up to 6 months
  Mortality
RRT Required | During course of ICU stay, could be up to 6 months
  Need for RRT

CONTACTS AND LOCATIONS:
Overall Officials: George F Alvarez, MD, Principal Investigator — Alberta Health services
Locations (2):
- Canada (2):
  - Peter Lougheed Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Once the results have been analyzed and published the de-identified data will be made available to other researchers
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available once published. It will be made available for 5 years as per University of Calgary data storage protocol.

REFERENCES:
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] Minasyan H. Sepsis and septic shock: Pathogenesis and treatment perspectives. J Crit Care. 2017 Aug;40:229-242. doi: 10.1016/j.jcrc.2017.04.015. Epub 2017 Apr 18. PMID 28448952
- [Background] Fisher CJ Jr, Dhainaut JF, Opal SM, Pribble JP, Balk RA, Slotman GJ, Iberti TJ, Rackow EC, Shapiro MJ, Greenman RL, et al. Recombinant human interleukin 1 receptor antagonist in the treatment of patients with sepsis syndrome. Results from a randomized, double-blind, placebo-controlled trial. Phase III rhIL-1ra Sepsis Syndrome Study Group. JAMA. 1994 Jun 15;271(23):1836-43. PMID 8196140
- [Background] Cohen J, Carlet J. INTERSEPT: an international, multicenter, placebo-controlled trial of monoclonal antibody to human tumor necrosis factor-alpha in patients with sepsis. International Sepsis Trial Study Group. Crit Care Med. 1996 Sep;24(9):1431-40. doi: 10.1097/00003246-199609000-00002. PMID 8797612
- [Background] Abraham E, Reinhart K, Opal S, Demeyer I, Doig C, Rodriguez AL, Beale R, Svoboda P, Laterre PF, Simon S, Light B, Spapen H, Stone J, Seibert A, Peckelsen C, De Deyne C, Postier R, Pettila V, Sprung CL, Artigas A, Percell SR, Shu V, Zwingelstein C, Tobias J, Poole L, Stolzenbach JC, Creasey AA; OPTIMIST Trial Study Group. Efficacy and safety of tifacogin (recombinant tissue factor pathway inhibitor) in severe sepsis: a randomized controlled trial. JAMA. 2003 Jul 9;290(2):238-47. doi: 10.1001/jama.290.2.238. PMID 12851279
- [Background] Afshari A, Wetterslev J, Brok J, Moller A. Antithrombin III in critically ill patients: systematic review with meta-analysis and trial sequential analysis. BMJ. 2007 Dec 15;335(7632):1248-51. doi: 10.1136/bmj.39398.682500.25. Epub 2007 Nov 23. PMID 18037615
- [Background] Ranieri VM, Thompson BT, Barie PS, Dhainaut JF, Douglas IS, Finfer S, Gardlund B, Marshall JC, Rhodes A, Artigas A, Payen D, Tenhunen J, Al-Khalidi HR, Thompson V, Janes J, Macias WL, Vangerow B, Williams MD; PROWESS-SHOCK Study Group. Drotrecogin alfa (activated) in adults with septic shock. N Engl J Med. 2012 May 31;366(22):2055-64. doi: 10.1056/NEJMoa1202290. Epub 2012 May 22. PMID 22616830
- [Background] Santacruz CA, Pereira AJ, Celis E, Vincent JL. Which Multicenter Randomized Controlled Trials in Critical Care Medicine Have Shown Reduced Mortality? A Systematic Review. Crit Care Med. 2019 Dec;47(12):1680-1691. doi: 10.1097/CCM.0000000000004000. PMID 31567349
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] van der Meche FG, Schmitz PI. A randomized trial comparing intravenous immune globulin and plasma exchange in Guillain-Barre syndrome. Dutch Guillain-Barre Study Group. N Engl J Med. 1992 Apr 23;326(17):1123-9. doi: 10.1056/NEJM199204233261705. PMID 1552913
- [Background] Barth D, Nabavi Nouri M, Ng E, Nwe P, Bril V. Comparison of IVIg and PLEX in patients with myasthenia gravis. Neurology. 2011 Jun 7;76(23):2017-23. doi: 10.1212/WNL.0b013e31821e5505. Epub 2011 May 11. PMID 21562253
- [Background] Mandawat A, Kaminski HJ, Cutter G, Katirji B, Alshekhlee A. Comparative analysis of therapeutic options used for myasthenia gravis. Ann Neurol. 2010 Dec;68(6):797-805. doi: 10.1002/ana.22139. PMID 21061395
- [Background] Bonnan M, Cabre P. Plasma exchange in severe attacks of neuromyelitis optica. Mult Scler Int. 2012;2012:787630. doi: 10.1155/2012/787630. Epub 2012 Feb 12. PMID 22474589
- [Background] DeSena AD, Noland DK, Matevosyan K, King K, Phillips L, Qureshi SS, Greenberg BM, Graves D. Intravenous methylprednisolone versus therapeutic plasma exchange for treatment of anti-N-methyl-D-aspartate receptor antibody encephalitis: A retrospective review. J Clin Apher. 2015 Aug;30(4):212-6. doi: 10.1002/jca.21363. Epub 2015 Feb 9. PMID 25664728
- [Background] Rock GA, Shumak KH, Buskard NA, Blanchette VS, Kelton JG, Nair RC, Spasoff RA. Comparison of plasma exchange with plasma infusion in the treatment of thrombotic thrombocytopenic purpura. Canadian Apheresis Study Group. N Engl J Med. 1991 Aug 8;325(6):393-7. doi: 10.1056/NEJM199108083250604. PMID 2062330
- [Background] Sarode R, Bandarenko N, Brecher ME, Kiss JE, Marques MB, Szczepiorkowski ZM, Winters JL. Thrombotic thrombocytopenic purpura: 2012 American Society for Apheresis (ASFA) consensus conference on classification, diagnosis, management, and future research. J Clin Apher. 2014 Jun;29(3):148-67. doi: 10.1002/jca.21302. Epub 2013 Oct 17. PMID 24136342
- [Background] Reeves JH. A review of plasma exchange in sepsis. Blood Purif. 2002;20(3):282-8. doi: 10.1159/000047021. PMID 11867876
- [Background] Zhou F, Peng Z, Murugan R, Kellum JA. Blood purification and mortality in sepsis: a meta-analysis of randomized trials. Crit Care Med. 2013 Sep;41(9):2209-20. doi: 10.1097/CCM.0b013e31828cf412. PMID 23860248
- [Background] Scharfman WB, Tillotson JR, Taft EG, Wright E. Plasmapheresis for meningococcemia with disseminated intravascular coagulation. N Engl J Med. 1979 May 31;300(22):1277-8. No abstract available. PMID 431695
- [Background] Vain NE, Mazlumian JR, Swarner OW, Cha CC. Role of exchange transfusion in the treatment of severe septicemia. Pediatrics. 1980 Nov;66(5):693-7. PMID 7432874
- [Background] Bjorvatn B, Bjertnaes L, Fadnes HO, Flaegstad T, Gutteberg TJ, Kristiansen BE, Pape J, Rekvig OP, Osterud B, Aanderud L. Meningococcal septicaemia treated with combined plasmapheresis and leucapheresis or with blood exchange. Br Med J (Clin Res Ed). 1984 Feb 11;288(6415):439-41. doi: 10.1136/bmj.288.6415.439. PMID 6419956
- [Background] Lercari G, Paganini G, Malfanti L, Rolla D, Machi AM, Rizzo F, Cannella G, Valbonesi M. Apheresis for severe malaria complicated by cerebral malaria, acute respiratory distress syndrome, acute renal failure, and disseminated intravascular coagulation. J Clin Apher. 1992;7(2):93-6. doi: 10.1002/jca.2920070211. PMID 1429495
- [Background] Gardlund B, Sjolin J, Nilsson A, Roll M, Wickerts CJ, Wikstrom B, Wretlind B. Plasmapheresis in the treatment of primary septic shock in humans. Scand J Infect Dis. 1993;25(6):757-61. doi: 10.3109/00365549309008575. PMID 8052817
- [Background] Busund R, Koukline V, Utrobin U, Nedashkovsky E. Plasmapheresis in severe sepsis and septic shock: a prospective, randomised, controlled trial. Intensive Care Med. 2002 Oct;28(10):1434-9. doi: 10.1007/s00134-002-1410-7. Epub 2002 Jul 23. PMID 12373468
- [Background] Long EJ, Taylor A, Delzoppo C, Shann F, Pearson G, Buckley D, Butt W. A randomised controlled trial of plasma filtration in severe paediatric sepsis. Crit Care Resusc. 2013 Sep;15(3):198-204. PMID 23944206
- [Background] Nguyen TC, Han YY, Kiss JE, Hall MW, Hassett AC, Jaffe R, Orr RA, Janosky J, Carcillo JA. Intensive plasma exchange increases a disintegrin and metalloprotease with thrombospondin motifs-13 activity and reverses organ dysfunction in children with thrombocytopenia-associated multiple organ failure. Crit Care Med. 2008 Oct;36(10):2878-87. doi: 10.1097/ccm.0b013e318186aa49. PMID 18828196
- [Background] Reeves JH, Butt WW, Shann F, Layton JE, Stewart A, Waring PM, Presneill JJ. Continuous plasmafiltration in sepsis syndrome. Plasmafiltration in Sepsis Study Group. Crit Care Med. 1999 Oct;27(10):2096-104. doi: 10.1097/00003246-199910000-00003. PMID 10548188
- [Background] Knaup H, Stahl K, Schmidt BMW, Idowu TO, Busch M, Wiesner O, Welte T, Haller H, Kielstein JT, Hoeper MM, David S. Early therapeutic plasma exchange in septic shock: a prospective open-label nonrandomized pilot study focusing on safety, hemodynamics, vascular barrier function, and biologic markers. Crit Care. 2018 Oct 30;22(1):285. doi: 10.1186/s13054-018-2220-9. PMID 30373638
- [Background] Szczepiorkowski ZM, Winters JL, Bandarenko N, Kim HC, Linenberger ML, Marques MB, Sarode R, Schwartz J, Weinstein R, Shaz BH; Apheresis Applications Committee of the American Society for Apheresis. Guidelines on the use of therapeutic apheresis in clinical practice--evidence-based approach from the Apheresis Applications Committee of the American Society for Apheresis. J Clin Apher. 2010;25(3):83-177. doi: 10.1002/jca.20240. PMID 20568098